#### **TITLE PAGE**

**Protocol Number:** C-17-TS13

**Protocol Title:** Clinical Study to Evaluate the Performance the truSculpt

Radiofrequency Device for Lipolysis of Abdominal Fat

**Sponsor:** Cutera, Inc.

3240 Bayshore Boulevard

Brisbane, CA 94005



Principal Investigator: Stephen Ronan, MD



**Version, Date:** Version 2, Dated July 6, 2017

## **Statement of Compliance**

The study will be conducted in accordance with the design and specific provisions of this IRB approved protocol, in accordance with the ethical principles that have their origin in the Declaration of Helsinki, and that are consistent with Good Clinical Practice (GCP) and the applicable regulatory requirement(s).

**NOTE:** The confidential information in the following document is provided to you as an Investigator, potential Investigator, or consultant for review by you, your staff, and applicable Institutional Review Board. By accepting this document, you agree that the information contained herein will not be disclosed to others, without written authorization from Cutera, Inc. except to the extent necessary to obtain informed consent from those persons to whom the device will be administered.

## Protocol Signature Page - Principal Investigator

## PROTOCOL C-17-TS13

Study Title: Clinical Study to Evaluate the Performance the truSculpt Radiofrequency Device for

**Lipolysis of Abdominal Fat** 

## Protocol Version 2.0, Dated July 06, 2017

I have received and read the protocol dated July 06, 2017 and agree to adhere to the requirements. I am aware that my adherence to the above protocol is mandatory and that any changes in the protocol or informed consent form must first be approved by Cutera, Inc. and the Institutional Review Board, except those changes necessary to eliminate apparent immediate hazards to subjects. I will provide copies of this protocol and all pertinent information to the study personnel under my supervision. I will discuss this material with them and ensure they are fully informed regarding their role in the study. I will ensure that the study is conducted in compliance with the protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements, and with the reviewing Institutional Review Board (IRB) requirements. I agree to commence this study only after documented IRB approval is obtained.

Principal Investigator

Signature

STEPHEN KONAN, MD

Date

# **Table of Contents**

| Proto | col Su | mmary | 5 |
|---|---|---|---|
| 1 F | URPC | OSE | 6 |
| 2 E | BACKE | ROUND INFORMATION | 6 |
| 3 S | TUDY | OBJECTIVES | 7 |
| 4 S | TUDY | DESIGN | 7 |
| 4 | 1.1.1 | Efficacy endpoints | 7 |
| 4 | 1.1.2 | Safety Endpoint | 7 |
| 4.2 | Sti | udy Duration | 8 |
| 4.3 | Sti | udy Assessments | 8 |
| 4 | l.3.1 | Safety Assessments | 8 |
| 4.4 | Sti | udy Discontinuation | 8 |
| 4.5 | Inv | vestigator Selection | 8 |
| 5 S | TUDY | POPULATION | 8 |
| 5.1 | St | udy Subject Recruitment and Selection | 8 |
| 5 | 5.1.1 | Inclusion Criteria | 9 |
| 5 | 5.1.2 | Exclusion Criteria | 9 |
| 5.2 | Su | bject Numbering | 10 |
| 5.3 | Su | bject Discontinuation Criteria | 10 |
| 6 S | TUDY | PROCEDURES | 10 |
| 6.1 | Sc | reening and Enrollment Visit Procedures | 10 |
| 6.2 | RF | Treatment Visit | 10 |
| 6.3 | Bio | ppsy Collection Visit | 11 |
| 7 <i>P</i> | ADVER | RSE DEVICE EFFECTS | 12 |
| 7.1 | De | finitions | 12 |
| 7 | 7.1.1 | Adverse Device Effect (ADE) | 12 |
| 7 | 7.1.2 | Serious Adverse Device Effect (SADE) | 12 |
| 7 | 7.1.3 | Anticipated Serious Adverse Device Effect (ASADE) | 12 |
| 7 | 7.1.4 | Unanticipated Serious Adverse Device Effect (USADE/UADE) | 12 |
| 7.2 | | cording Adverse Device Effects | |
| 7.3 | Fo | llow-up of Subjects after ADEs | 14 |
| 8 F | | ITIAL RISKS / BENEFITS | |
| 8.1 | Ро | tential Risks | 14 |
| 8.2 | Po | tential Benefits | 15 |

| ; | 3.3 | Risk Management | 15 |
|----|--------|----------------------------------------------|----|
| 9 | DAT | A ANALYSIS PLAN | 16 |
| 9 | 9.1 | Sample Size | 16 |
| 9 | 9.2 | Analysis Sets | 16 |
| 9 | 9.3 | Analysis of Efficacy Endpoints | 16 |
| | 9.3. | 1 Primary Endpoint Analysis | 16 |
| 9 | 9.4 | Safety Analyses | 16 |
| 10 | SUB | JECT PAYMENT | 16 |
| 11 | STU | DY MANAGEMENT AND ADMINISTRATIVE PROCEDURES | 16 |
| : | 11.1 | Training and Monitoring | 16 |
| | 11.2 | Informed Consent | 17 |
| | 11.3 | Protocol Compliance | 17 |
| | 11.3.1 | Protocol Amendments | 17 |
| | 11.3.2 | Protocol Deviations | 17 |
| | 11.4 | Study Personnel | 18 |
| | 11.5 | Disclosure of Financial Interest | 18 |
| | 11.6 | Data Collection, Record Keeping and Storage | 18 |
| | 11.7 | Subject Confidentiality | 19 |
| | 11.8 | Publication Policy | 20 |
| RE | FERE | ENCES | 21 |
| Ар | pendi | x 1: Study Schedule | 23 |
| Ap | pendi | x 2: Pain Rating Scale | 24 |
| Ар | pendi | x 3: Fitzpatrick Skin Type Classification | 25 |
| αA | pendi | x 4: Before and After Treatment Instructions | 26 |

# **Protocol Summary**

| Title | Clinical Study to Evaluate the Performance the truSculpt<br>Radiofrequency Device for Lipolysis of Abdominal Fat |
|---|---|
| Objective | To evaluate the truSculpt Radiofrequency Device for non-<br>invasive fat reduction in abdominal tissue |
| Study Design | A single-center, prospective, non-randomized, open-label study |
| Enrollment | Approximately 14 subjects |
| Primary Endpoint | Histological evaluation of tissue for selective fat necrosis, with sparing of the dermis and epidermis, following truSculpt treatment vs. untreated contralateral control |
| Safety Endpoint | Incidence and severity of adverse device effects during the study period, including subject pain level during RF treatment |
| Subject Population | Female and male subjects, age 24 to 60 years, Fitzpatrick skin type I-VI |
| Planned Schedule | First subject enrolled: June 2017 |
| | Last subject last visit: June 2018 |

  Version 2.0,06JUL 2017

#### 1 PURPOSE

The purpose of this investigation is to evaluate the performance of the truSculpt Radiofrequency Device for non-invasive lipolysis of abdominal fat.

#### 2 BACKGROUND INFORMATION

Unwanted excess fat pockets/bulges have been among the top concerns expressed by patients in the aesthetic field. Although surgical interventions produce the most definitive results with body contouring, these invasive methods require significant recovery time and come with inherent risks.

As a non-invasive option, laser, intense pulsed light (IPL), RF, or a combination of these technologies have been developed to reduce cellulite and body circumference with minimal recovery time and risks [1]. The tightening effect of the thermal energy generated by these devices has been used for reduction in cellulite and body circumference in areas including but not limited to arms, abdomen, thigh, back and flanks [2-14]. Although lasers and IPLs can target the deep dermal layers, the thermal effects of these devices are limited due to light scattering and energy absorption by water in the dermis.

RF, which is the most studied device in the non-ablative category, uses electrical current rather than light energy. Unlike light energy, radio waves can penetrate deeper depending on the frequency of operation. RF can be used with all Fitzpatrick skin types without jeopardizing epidermal integrity [15].




Sample labeling and directions for use can be found in the Operator's Manual for this device.

| Table 1. truSculpt RF Device Specifications |
|---------------------------------------------|
| RF Power |
| Pulse Duration |
| Frequency |
| Target Skin Temperature |
| Handpiece Size |

#### 3 STUDY OBJECTIVES

The objective of this study is to evaluate the truSculpt Radiofrequency Device for non-invasive fat reduction in abdominal tissue.

#### 4 STUDY DESIGN

This is a single-center, prospective, non-randomized, open-labeled study in approximately 14 subjects, age 24 to 60 years, who are scheduled for abdominoplasty, and will undergo one RF treatment in the abdominal region. Subjects will receive 1 RF treatment with the truSculpt device

One treatment will be performed by the truSculpt device on one abdominal subarea, while the other abdominal subarea will not be treated and will serve as a control. Subjects will have incisional or full-thickness punch skin biopsies. Biopsies will be harvested from tissue to be removed during the abdominoplasty, and will subsequently be cultured. At least two biopsy samples for each subject will be obtained during the abdominoplasty: at least one from the treatment area and at least one from the control area. The purpose of the biopsies is to examine and compare potential histological changes in cutaneous and sub-cutaneous tissue levels that occur as a result of RF treatment.

#### 4.1 Study Endpoints

#### 4.1.1 Efficacy endpoints

## 4.1.1.1 Primary Efficacy Endpoint

 Histological evaluation of tissue for selective fat necrosis, with sparing of the dermis and epidermis, following truSculpt treatment vs. untreated bilateral control.

#### 4.1.2 Safety Endpoint

 Incidence and severity of adverse device effects during the study period, including subject pain level during RF treatment.


#### 4.2 Study Duration

Subjects enrolled in this trial will be asked to participate for up to 3 months and will complete 3 visits: 1 screening visit, 1 RF treatment visit, and 1 follow-up visit (biopsy collection visit) on the day of their planned abdominoplasty surgery.

## 4.3 Study Assessments

## 4.3.1 Safety Assessments

## 4.3.1.1 Incidence and Severity of Adverse Events:

Following the first RF treatment, adverse device effects (ADEs) will be assessed post-treatment and at each subsequent subject visit using the following scale:

- 1= mild: requires minimal or no treatment and does not interfere with the Subject's daily activities.
- 2= moderate: may cause some interference with functioning.
- 3= severe: interrupts Subject's usual daily activity and may require treatment.

## 4.3.1.2 Treatment-related Discomfort

Subjects will be asked to rate the average amount of discomfort experienced during RF treatment using the Pain Rating Scale found in Appendix 3.

## 4.4 Study Discontinuation

The study sponsor has the right to terminate this study at any time. Reasons for terminating the study may include, but are not limited to, unsatisfactory subject enrollment or the incidence or severity of adverse events in this study, or other studies with the study device, indicates a potential health hazard to subjects.

#### 4.5 Investigator Selection

Investigators will be invited to participate in the study based on their medical specialty, experience conducting clinical research studies and experience in the use of energy based devices for aesthetic indications. The site's access to potential study subjects and ability to cooperate with study requirements will also be considered.

#### 5 STUDY POPULATION

## 5.1 Study Subject Recruitment and Selection

Approximately 14 male or female subjects, ages 24 to 60, Fitzpatrick Skin Type I-VI, who are scheduled for abdominoplasty, and will undergo one RF treatment on tissue to be removed during their abdominoplasty, will be studied. Subjects will be recruited to participate from those patients who present themselves to the site requesting abdominoplasty surgery, or from those patients who respond to advertisement. Only subjects who meet all Inclusion and Exclusion Criteria and provide written informed consent will be enrolled into the study.

Each subject will be evaluated by the Investigator to assess his/her suitability for entry into the study according to the following inclusion and exclusion criteria.


## 5.1.1 Inclusion Criteria

To be included in the study, subjects must meet all of the following Inclusion Criteria:

| 1. | Male or Female, 24 to 60 years of age (inclusive) |
|---|---|
| 2. | Fitzpatrick Skin Type I – VI (Appendix 3) |
| 3. | Has visible fat bulges or skin laxity in the abdominal region |
| 4. | Scheduled to undergo surgery (abdominoplasty). |
| 5. | Non-smoking for at least 6 months and willing to refrain from smoking for the duration |
| | of the study. |
| 6. | Subject must agree to not undergo any other procedure(s) in the abdominal region |
| | during the study period. |
| 7. | Subject must be able to read, understand and sign the Informed Consent Form. |
| 8. | Subject must adhere to the follow-up schedule and study instructions. |
| 9. Subject must adhere to the same diet/ exercise/medication regimen for th | |
| | course of the study. |
| 10. | Willing to provide histology samples during the surgery from the intended to be |
| harvested areas. | |
| 11. | Post-menopausal or surgically sterilized, or using a medically acceptable form of birth |
| | control at least 3 months prior to enrollment and during the entire course of the study, |
| | and no plans to become pregnant. |

## 5.1.2 Exclusion Criteria

Subjects will be excluded from the study if they meet any of the following Exclusion Criteria:

| <ol> <li>Participation in a clinical trial of another device or drug in the target area during the study period.</li> <li>Any type of prior cosmetic treatment to the target area within 12 months of study participation e.g., radiofrequency, cryolysis or light-based treatments.</li> <li>Any prior invasive cosmetic surgery to the target area, such as liposuction.</li> <li>Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant.</li> <li>Has metal implant(s) within the body, such as surgical clips, plates and screws, intrauterine device (IUD), artificial heart valves or artificial joints.</li> <li>Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders.</li> <li>Diagnosed or documented immune system disorders.</li> <li>Diagnosed or documented immune system disorders.</li> <li>History of any disease or condition that could impair wound healing.</li> <li>History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.</li> <li>History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area.</li> <li>Infection, dermatitis, rash or other skin abnormality in the target area.</li> <li>Currently undergoing systemic chemotherapy or radiation treatment for cancer, or</li> </ol> | | |
|---|---|---|
| participation e.g., radiofrequency, cryolysis or light-based treatments. 3. Any prior invasive cosmetic surgery to the target area, such as liposuction. 4. Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant. 5. Has metal implant(s) within the body, such as surgical clips, plates and screws, intrauterine device (IUD), artificial heart valves or artificial joints. 6. Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders. 7. Diagnosed or documented immune system disorders. 8. History of any disease or condition that could impair wound healing. 9. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen. 10. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area. 11. Infection, dermatitis, rash or other skin abnormality in the target area. | 1. | |
| <ol> <li>Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant.</li> <li>Has metal implant(s) within the body, such as surgical clips, plates and screws, intrauterine device (IUD), artificial heart valves or artificial joints.</li> <li>Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders.</li> <li>Diagnosed or documented immune system disorders.</li> <li>History of any disease or condition that could impair wound healing.</li> <li>History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.</li> <li>History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area.</li> <li>Infection, dermatitis, rash or other skin abnormality in the target area.</li> </ol> | 2. | , |
| stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant. 5. Has metal implant(s) within the body, such as surgical clips, plates and screws, intrauterine device (IUD), artificial heart valves or artificial joints. 6. Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders. 7. Diagnosed or documented immune system disorders. 8. History of any disease or condition that could impair wound healing. 9. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen. 10. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area. 11. Infection, dermatitis, rash or other skin abnormality in the target area. | 3. | Any prior invasive cosmetic surgery to the target area, such as liposuction. |
| <ul> <li>intrauterine device (IUD), artificial heart valves or artificial joints.</li> <li>6. Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders.</li> <li>7. Diagnosed or documented immune system disorders.</li> <li>8. History of any disease or condition that could impair wound healing.</li> <li>9. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.</li> <li>10. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area.</li> <li>11. Infection, dermatitis, rash or other skin abnormality in the target area.</li> </ul> | 4. | stimulator implant, cochlear implant or any other electronically, magnetically or |
| peripheral vascular disease or pertinent neurological disorders. 7. Diagnosed or documented immune system disorders. 8. History of any disease or condition that could impair wound healing. 9. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen. 10. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area. 11. Infection, dermatitis, rash or other skin abnormality in the target area. | 5. | |
| <ol> <li>History of any disease or condition that could impair wound healing.</li> <li>History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.</li> <li>History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area.</li> <li>Infection, dermatitis, rash or other skin abnormality in the target area.</li> </ol> | 6. | |
| <ol> <li>History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.</li> <li>History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area.</li> <li>Infection, dermatitis, rash or other skin abnormality in the target area.</li> </ol> | 7. | Diagnosed or documented immune system disorders. |
| area, unless treatment is conducted following a prophylactic regimen. 10. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area. 11. Infection, dermatitis, rash or other skin abnormality in the target area. | 8. | History of any disease or condition that could impair wound healing. |
| in the treatment area. 11. Infection, dermatitis, rash or other skin abnormality in the target area. | 9. | • |
| | 10. | , |
| 12. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or | 11. | Infection, dermatitis, rash or other skin abnormality in the target area. |
| | 12. | Currently undergoing systemic chemotherapy or radiation treatment for cancer, or |


| | history of treatment in the target area within 3 months of study participation. |
|---|---|
| 13. Pregnant or currently breastfeeding. | |
| 14. | As per the Investigator's discretion, any physical or mental condition which might make |
| it unsafe for the subject to participate in this study. | |

## 5.2 Subject Numbering

Each enrolled subject will be assigned a subject ID number, comprised of the sequential number assigned for each subject treated and the subject initials. The subject initials will be comprised of the first letter of the first and last name.

## 5.3 Subject Discontinuation Criteria

If possible, every subject should remain in the study until completion of the required follow-up period. However, participation in this study is completely voluntary and a subject can choose to withdraw from the study at any time. In addition, a subject can be discontinued for any of the following reasons: the Principal Investigator decides that continuing in the study would not be in the subject's best interest, a subject is noncompliant with the protocol, a subject has a serious reaction to the treatment, or the study is stopped. In addition, subjects may be discontinued from the study if s/he develops any of the exclusion criteria during the study period. A subject will be considered lost to follow-up only after three unsuccessful, documented attempts to contact the subject have been made.

#### **6 STUDY PROCEDURES**

A summary of all required study procedures and assessments can be found in Appendix 1.

## 6.1 Screening and Enrollment Visit Procedures

The following screening procedures will be performed:

- 1. Informed Consent process.
- 2. Review of subject medical history.
- 3. Assessment of treatment area.
- 4. Assessment of concomitant medications.
- 5. Assign subject to a subgroup.

#### 6.2 RF Treatment Visit

The following procedures will be performed at the RF Treatment Visit:

- 1. If needed, cleanse subject's treatment area with a mild cleanser to remove any cosmetics, perfume or lotions and then dry the area.
- 2. Prior to performing RF treatment, the Investigator should confirm the subject continues to meet the study eligibility criteria, including asking about any changes in medical history and/or concomitant medications or significant increase or decrease in subject weight.
- 3. Using a surgical marker, mark the subject's abdomen as it will be marked on the day of the subsequent planned abdominoplasty procedure.


- 4. Place the return pad on the subject's upper lateral back. Connect the neutral electrode cable after the return pad has been applied.
- 5. The subject should be lying down and comfortable while undergoing RF treatment and the operator should have easy access to the treatment area.
- Conduct RF treatment according to the parameters listed in Table 2 with one imprint applied to the subject's abdomen over the tissue intended to be removed during the following abdominoplasty procedure.

| Table 2. TruSculpt RF Device Treatment |
|----------------------------------------|
| RF Power |
| Pulse Duration |
| Frequency |
| Target Skin Temperature |
| Handpiece Size |

- 7. Place the handpiece on the skin of the area to be treated and ensure the electrode is in full contact with the skin at all times. Do not apply excess pressure as this may diminish treatment effects and cause additional subject discomfort. The operator must wear surgical gloves during RF treatment.
- 8. After the imprint is delivered, an image will be taken of the subject's markings and posttreatment hyperemia pattern showing the location of the imprint. The image will be added to the subject's chart. The pulse duration for the imprint and the target temperature achieved during RF treatment will be recorded in the subject's chart.
- 9. The subject will be asked to rate the average level of discomfort experienced during and after completion of treatment using the Pain Rating Scale found in Appendix 3.
- 10. Investigator will assess and record any immediate post-treatment adverse device effects.
- 11. The "Before and After Treatment Instructions" will be explained and provided to the subject (see Appendix 4).

## 6.3 Biopsy Collection Visit

The Biopsy Collection visit will occur on the same day as the abdominoplasty surgery. The following procedures will be performed prior to and during abdominoplasty surgery:

- 1. Review of subject medical history.
- 2. Assess and record any additions, changes and/or deletions in prescription and nonprescription concomitant medications since the previous study visit.
- 3. Record severity and duration of any adverse device effects following RF treatment and assess for any new adverse device effects.
- 4. Biopsy collection procedure:
  - a. Refer to the patient chart and identify the RF treatment location.
  - b. During the biopsy collection procedure, at least one skin biopsy (approximately 10 mm x 10 mm; full thickness) will be taken from the area treated with RF; and at least one skin biopsy (approximately 10 mm x 10 mm; full thickness) will be taken from an equivalent contralateral non-treated area as a control.


c. Each biopsy sample will be immediately placed in the prepared fixative vials, making sure the samples are fully submerged in the solution. The vials will be labeled with the subject ID number, subject initials and biopsy date. The vials will be randomly numbered, and the numbers of the vials containing the biopsy from the RF treated and control skin will be recorded in the patient chart. The histologist will remain blinded to the nature of each biopsy sample (treatment or control).

#### 7 FADVERSE DEVICE EFFECTS

#### 7.1 Definitions

## 7.1.1 Adverse Device Effect (ADE)

An adverse device effect (ADE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, device users or other persons, related to the investigational medical device. ADEs <u>may be previously identified</u> in nature, incidence, severity or outcome in the study protocol, informed consent document, device operator manual, other risk analysis documentation or regulatory application.

## 7.1.2 Serious Adverse Device Effect (SADE)

A serious adverse device effect (SADE) is any adverse device effect, related to the use of an investigational device or clinical study device, that:

- led to a death;
- led to a serious deterioration in the health of the subject that:
  - resulted in a life-threatening illness or injury;
  - resulted in a permanent impairment of a body structure or body function;
  - required in-patient hospitalization or prolongation of existing hospitalization;
  - resulted in medical or surgical intervention to prevent permanent impairment to a body structure or a body function
- led to fetal distress, fetal death or a congenital abnormality or birth defect.

## 7.1.3 Anticipated Serious Adverse Device Effect (ASADE)

An anticipated serious adverse device effect (ASADE) is any SADE on health or safety or any life-threatening problem or death caused by, or associated with the device, if that effect, problem, or death was previously identified in nature, severity, or degree of incidence in the investigational plan, informed consent, operator manual, other risk analysis documentation or regulatory application; or any other serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

#### 7.1.4 Unanticipated Serious Adverse Device Effect (USADE/UADE)

An unanticipated serious adverse device effect (USADE) is any SADE on health or safety or any life-threatening problem or death caused by, or associated with the device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, informed consent, operator manual, other risk analysis documentation, or regulatory application; or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.


"Clinical Study to Evaluate the Performance the TruSculpt Radiofrequency Device for Lipolysis of Abdominal Fat"

In subjects, the ADEs/SADEs include the effects related to the investigational medical device (clinical study device), the comparator or the procedures involved. For device users or other persons (other clinical staff in the treatment room) ADE/SADE is restricted to the effects related to investigational medical devices. ADEs/SADEs may include the effects (1) resulting from insufficient or inadequate instructions for use, deployment, installation, or operation, or any malfunction of the investigational medical device; or (2) resulting from user error or from intentional misuse of the investigational medical device.

**Adverse Event Occurrence** (i.e., Untoward Medical Occurrence) Is it device, comparator or procedure related? yes Adverse Device Event (ADE) no Does it meet - Reported on Visit CRF seriousness - Examples: erythema, edema, bruise, 1<sup>st</sup> and 2<sup>nd</sup> criteria? degree burn yes **Serious Adverse Device** Effect (SADE) yes **Unanticipated Serious Adverse Device Effect** no (USADE/UADE) Is it - Reported on Cutera SADE Form anticipated? - Reported on ADE CRF - Examples: seizure, event leading to death yes

Figure 1. Flowchart for classification of adverse device effects [19]

# **Anticipated Serious Adverse Device Effect** (ASADE)

- Reported on Cutera SADE Form
- Reported on ADE CRF
- Examples: 3<sup>rd</sup> degree burn, eye damage from laser

## 7.2 Recording Adverse Device Effects

All potential ADEs will be evaluated and must be recorded in the subject's medical chart and in the study case report forms. ADEs will be monitored and tracked from the time of the first RF treatment.

At each contact with the subject, the Investigator will seek information on ADEs by specific questioning and, as appropriate, by examination. ADEs may be observed by the Investigator and/or clinical research staff, elicited from the subject and/or family member or volunteered by the subject. All observed and volunteered adverse signs and symptoms (both expected and unexpected), regardless of severity or frequency, will be recorded in the case histories (medical chart and CRFs). Included in the description should be the nature of the sign or symptom, the date of onset, date of resolution (duration), the severity, whether the event was expected or unexpected (anticipated or unanticipated), the relationship to study treatment or other therapy, the action taken (if any), and the outcome.

All SADEs and UADEs must be reported according to Cutera and IRB requirements.

#### 7.3 Follow-up of Subjects after ADEs

All reported ADEs should be followed until resolution or until the subject's participation in the study ends. Resolutions of such events are to be documented on the appropriate CRF pages. All ADEs that result in permanent discontinuation from this clinical trial, whether serious or not, will also be reported on the Subject Non-Completion of Study Form.

## 8 POTENTIAL RISKS / BENEFITS

#### 8.1 Potential Risks

The known risks and adverse device effects associated with the study device or treatment procedure are shown in **Table 3**.

Table 3. Potential Study Risks

| Table 3. Potential Study Risks or ADEs/SADEs | | | |
|---|---|---|---|
| STUDY DEVICE/PROCEDURE RELATED | | | |
| Type of Adverse Device Effect | Severity | Expected<br>Duration | Frequency |
| Abrasion | Mild to Severe | 3-14 days | Very Rare |
| Bleeding | Mild | Up to 1 hour | Very Rare |
| Blanching | Mild | > 24 hours | Very Rare |
| Blistering | Mild to Severe | 1-14 days | Rare |
| Burn | Moderate | 1-3 weeks | Rare |
| Contour Abnormalities/Cutaneous<br>Depressions | Mild to Severe | > 1 month | Uncommon |


| | 1 | 1 | |
|---|---|---|---|
| Crusting/Scabbing | Mild to Severe | 3-14 days | Rare |
| Edema (Swelling) | Mild to<br>Moderate | < 72 hours | Very Common |
| Erythema (Redness) | Mild to<br>Moderate | < 24 hours | Very Common |
| Hyperpigmentation | Mild to Severe | > 1 month | Rare |
| Hypopigmentation | Mild to Severe | > 1 month | Very Rare |
| Infection | Mild to Severe | 2-14 days | Rare |
| Palpable nodules | Mild to<br>Moderate | > 1 month | Common |
| Oozing | Mild to Severe | 2-14 days | Very Rare |
| Pain (Discomfort) | Mild to Severe | During procedure | Very Common |
| Purpura (Bruising) | Mild to<br>Moderate | 7-21 days | Common |
| Scarring | Mild to Severe | > 1 month | Rare |
| Textural Changes | Mild to Severe | > 1 month | Rare |
| Partial, over treatment, and/or no treatment with the study device(s) due to equipment problem (device malfunction) | Mild to Severe | | Rare |
| Improper treatment (partial, over-<br>treatment, and/or no treatment) with the<br>study device(s) due to user error | Mild to Severe | | Rare |
| Unintended injury to subject, user or others due to user error (e.g., unintentional treatment to non-target location) | Mild to Severe | | Rare |

#### 8.2 Potential Benefits

The subjects may or may not benefit from the treatment. Potential benefits include improved appearance of the treated abdominal and flank region and circumferential reduction in the treated abdominal and flank region. There is no guarantee of success.

## 8.3 Risk Management

The Investigator chosen for this study will have extensive and safe experience with the use of RF systems in dermatology applications. This is the most critical element in managing subject risk. In addition, the Investigators will be trained on the use of the Cutera RF device and any investigational handpieces.


#### 9 DATA ANALYSIS PLAN

## 9.1 Sample Size

The planned sample size of up to approximately 14 subjects was determined based on clinical judgement to provide sufficient information to evaluate the performance of RF treatment for lipolysis of abdominal fat.

#### 9.2 Analysis Sets

The efficacy analysis set will include all enrolled subjects who complete the RF treatment session using the study device.

The safety analysis set will include all subjects enrolled in the study who start the RF treatment session using the study device.

Missing data will not be imputed for efficacy or safety endpoints.

## 9.3 Analysis of Efficacy Endpoints

## 9.3.1 Primary Endpoint Analysis

Formal hypothesis testing and statistical analysis are not planned for this study. The primary efficacy endpoint data will be summarized descriptively for the control and treatment areas.

## 9.4 Safety Analyses

Device-related and procedure-related adverse effects (AEs) and subjects who prematurely terminate from the study due to an adverse device effect, including the treatment-related pain ratings, will be tabulated and analyzed. For a given AE term, counting will be done by subject, not by event, i.e. for a subject reporting the same AE more than once; the event will be counted only once, at the most severe and longest duration. The number and percentage of subjects experiencing each AE Term will be descriptively summarized. Subject pain ratings during treatment will also be summarized descriptively.

#### 10 SUBJECT PAYMENT

#### 11 STUDY MANAGEMENT AND ADMINISTRATIVE PROCEDURES

#### 11.1 Training and Monitoring

The investigators and site research staff will be trained on the study procedures. Sponsor representative(s) may be present at the site during the treatments to ensure that all procedures and documentation are in place.

Investigator will allow sponsor representatives to periodically review the study documentation. Monitoring of the site will occur at regular intervals to evaluate the progress of the study, verify the accuracy and completeness of CRFs against subject source documentation, assure that all protocol requirements, applicable FDA regulations and the investigator's obligations are being fulfilled and resolve any inconsistencies in the study records.


#### 11.2 Informed Consent

The investigator is responsible for ensuring that written informed consent, using an Institutional Review Board (IRB) approved informed consent document, is obtained from each subject before the performance of any protocol procedures, including administration of the study device. The informed consent document must comply with all essential elements as defined in 21 CFR 50.25 "Elements of Informed Consent" and must contain a statement that consent is freely given, the study involves research, the subject is aware of the risks and benefits of entering the study, and that the subject is free to withdraw from the study at any time. An evaluation of each candidate will be conducted by the investigator. Upon determining a subject's eligibility status, the subject will be offered the opportunity to participate in the study.

The investigator or the investigator's designee will inform all subjects regarding the purpose of the study and expected duration, as well as the potential risks and benefits that may result from participation. The subjects shall be informed by the investigator or investigator's designee that they are free to refuse participation in this clinical study. If they elect to participate, it will be made clear that they may withdraw from the study at any time without prejudicing further care.

The subjects will also be informed of alternative methods of treatment should they not wish to participate in the study.

The subjects will be given the opportunity to discuss the procedure, risks, benefits, alternative therapies, and the study requirements with the investigator and have any and all questions answered to the subjects' satisfaction. A signed and dated informed consent form must be obtained from the subject by the Investigator or the Investigator's designee prior to a subject's involvement in the study.

The acquisition of informed consent will be documented in the subject's medical records, as required by 21 CFR 812.140. A copy of the consent form will be given to the subject. The original consent forms will be kept in the CRF binder by the investigator and will be subject to review by Cutera or a representative of Cutera, and by appropriate regulatory bodies.

#### 11.3 Protocol Compliance

The principal investigator must comply with all terms of the protocol.

#### 11.3.1 Protocol Amendments

Neither the principal investigator nor the sponsor will modify or alter this protocol without first obtaining the concurrence of the other party (with the exception of amendments which involves mitigating a medical emergency or immediate health risk to the subject). The party initiating an amendment must confirm it clearly in writing and it must be signed and dated by the sponsor and the principal investigator. IRB approval must be obtained before implementation of an amendment.

#### 11.3.2 Protocol Deviations

All protocol deviations must be clearly described on the case report form (i.e., Cutera Protocol Deviation Form). Deviations from the protocol may include but are not limited to subject's failure to attend scheduled visit during a visit window, use of out of range treatment parameters and incomplete or


incorrect study procedures. Any medical emergency or immediate health risk to the subject which results in a protocol deviation and must be reported to the sponsor within 5 working days

Significant protocol deviations must be reported to IRB according to their policies.

#### 11.4 Study Personnel

Prior to the start of the study, the investigator must supply the sponsor with a list of the names and curricula vitae that describe the professional backgrounds of the clinically responsible study investigators (principal, sub-investigators), research nurses, and other possible participants (e.g. medical doctor, nurse, etc.).

#### 11.5 Disclosure of Financial Interest

Each investigator [principal and sub-investigator(s)] is required to disclose sufficient accurate financial information to the sponsor, to allow sponsor to submit complete and accurate certification or disclosure statements.

## 11.6 Data Collection, Record Keeping and Storage

The principal investigator is responsible for assuring that all study records including case report forms (CRFs), informed consent forms, device accountability records, source documents (e.g., medical records, histology reports etc.) and other study records are complete, accurate and recorded in a timely manner.

CRFs should not be the only record of a patient's participation in the study and will be used for transcribing data from source documents which are the point of first entry of data collected for each subject (with the exception of documents listed under **B**). The investigator or research staff at the site will ensure that:

## A. Source documentation thoroughly and adequately documents:

- 1. That patient is participating in a clinical study and has been properly informed and consented prior to participation in the study,
- 2. Medical history,
- 3. Concomitant medications,
- 4. Patient's condition upon entering and during the course of the study,
- 5. Any adverse event(s) that might have occurred (in addition to the Visit CRFs and/or Adverse Device Effect CRF and/or Cutera SADE form completed),
- 6. Results of any diagnostic tests/histology conducted during the study.

## B. The following data will be recorded directly onto CRFs:

- 7. Patient meets study inclusion and exclusion criteria,
- A record of the treatment parameters, including the date of each RF treatment and any other
  adjunct therapy, a drawing of the patients abdomen showing the treatment location, and the
  vial numbers containing control and treatment biopsies,
- 9. Any protocol deviations,
- 10. Subject Questionnaire(s),
- 11. Study related improvement assessments by the investigator or investigator's designee,


## 12. Treatment-related pain ratings.

## C. The following documents will be maintained in the study records:

- 13. The Investigator or the research staff will check signed informed consent for accuracy and will always keep the original copy of the signed informed consent in the CRF binder.
- 14. All correspondence with an Institutional Review Board (IRB), the sponsor, or FDA including required reports will also be retained in the study records.
- 15. Records of receipt, use or disposition of the investigational device.

All data entries on the CRFs will be recorded completely, promptly, and legibly using blue or black indelible ink pen and accuracy will be ensured. The corrections on CRFs will be made only by the investigator or the documented investigator's designee. To make a correction to an entry, the data will be crossed through with a single line (the original entry should be visible) and then will be initialed and dated by the person making the correction.

The study records will be maintained in a secure location throughout the duration of the study. Upon study completion or termination, records will be kept at a secure location until at least 2 years after the last approval of a marketing application and until there are no pending or contemplated marketing applications or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product.

## 11.7 Subject Confidentiality

This study preserves the confidentiality of all subjects under the Health Insurance Portability and Accountability Act of 1996 (HIPAA) Privacy Rule. The following safeguards will be in place to protect the privacy of the individuals who are the subjects of the health information to be used in the research and the confidentiality of that information:

The subjects will be informed by the investigator or the investigator's designee that their medical records will be kept as confidential as possible but may be subject to review by: (1) Cutera, or its representative; (2) reviewing IRB; and/or (3) by appropriate regulatory bodies (e.g. the US Food and Drug Administration (FDA), Department of Health and Human Services (DHHS) agencies).

Only pieces of personal information required for purposes of the study will be collected. The personal information will be collected and used to ensure subject eligibility for study participation, to conduct the study and to assess the results of the study as required and permitted by law. Subjects have the right to see and copy any of the information gathered about them and request changes if the information is not correct, until it is no longer kept by the investigator. Permission to use or disclose personal information, except for that has been collected and relied on may be cancelled by the subject by written notice. If the subject is withdrawn from the study, the information collected to that time may still be used to preserve the scientific integrity of the study. There is no expiration date to this authorization.

Subjects' identities will be kept confidential. Subjects will be assigned a unique study code that will not reveal the subjects' identity, and this code will be used on all study documents. To protect subject identity with regards to the photographs taken of the treatment areas, care will be taken to cover areas of photographs to protect identity. Techniques such as covering of eyes on full face photographs,


cropping off portions of the face in close-up photos will be used to obscure identifying characteristics in photographs. The results of research, including photographs, may be published in scientific journals, presented at medical meetings, and used in training and marketing materials but subject identities will not be disclosed.

## 11.8 Publication Policy

The investigator shall have the right to publish the results of the study. Unless mutually agreed upon in writing, prior to submission for publication of any manuscript, poster, presentation, abstract or other written or oral material describing the results of the study, the investigator shall allow sponsor to review manuscript, poster presentation, abstract or other written or oral material which describes the results of the study for the purpose only of determining if any patentable information is disclosed. At the sponsor's request, the investigator shall withhold any publication or presentation to permit sponsor to seek patent protection and to remove any confidential information from all publications.

The International Committee of Medical Journal Editors (ICMJE) member journals have adopted a trials registration policy as a condition for publication. This policy requires that all clinical trials be registered in a public trials registry such as ClinicalTrials.gov, which is sponsored by the National Library of Medicine. It is the responsibility of the sponsor to register this trial in ClinicalTrials.gov. Any clinical trial starting enrollment after September 27, 2007 must be registered either on or before the onset of patient enrollment.


#### REFERENCES

- 1. Ross EV, Yashar SS, Naseef GS, Barnette DJ, Skrobal M, Grevelink J, Anderson RR. A pilot study of in vivo immediate tissue contraction with CO2 skin laser resurfacing in a live farm pig. Dermatol Surg. 1999 Nov;25(11):851-6. PubMed PMID: 10594596.
- 2. Kulick M. Evaluation of the combination of radio frequency, infrared energy and mechanical rollers with suction to improve skin surface irregularities (cellulite) in a limited treatment area. J Cosmet Laser Ther. 2006 Dec;8(4):185-90. PubMed PMID: 19839171.
- 3. Alexiades-Armenakas M, Dover JS, Arndt KA. Unipolar radiofrequency treatment to improve the appearance of cellulite. J Cosmet Laser Ther. 2008 Sep;10(3):148-53. PubMed PMID: 18788033.
- 4. Sadick N. Tissue tightening technologies: fact or fiction. Aesthet Surg J. 2008 Mar-Apr;28(2):180-8. Review. PubMed PMID: 19083525.
- 5. Sukal SA, Geronemus RG. Thermage: the nonablative radiofrequency for rejuvenation. Clin Dermatol. 2008 Nov-Dec;26(6):602-7. PubMed PMID: 18940540.
- Elsaie ML. Cutaneous remodeling and photorejuvenation using radiofrequency devices. Indian J Dermatol. 2009 Jul;54(3):201-5. PubMed PMID: 20161847; PubMed Central PMCID: PMC2810682.
- 7. Emilia del Pino M, Rosado RH, Azuela A, Graciela Guzmán M, Argüelles D, Rodríguez C, Rosado GM. Effect of controlled volumetric tissue heating with radiofrequency on cellulite and the subcutaneous tissue of the buttocks and thighs. J Drugs Dermatol. 2006 Sep;5(8):714-22. PubMed PMID: 16989185.
- 8. Goldberg DJ, Fazeli A, Berlin AL. Clinical, laboratory, and MRI analysis of cellulite treatment with a unipolar radiofrequency device. Dermatol Surg. 2008 Feb;34(2):204-9; discussion 209. Epub 2007 Dec 17. PubMed PMID: 18093200.
- 9. Nootheti PK, Magpantay A, Yosowitz G, Calderon S, Goldman MP. A single center, randomized, comparative, prospective clinical study to determine the efficacy of the VelaSmooth system versus the Triactive system for the treatment of cellulite. Lasers Surg Med. 2006 Dec;38(10):908-12. PubMed PMID: 17163477.
- 10. Montesi G, Calvieri S, Balzani A, Gold MH. Bipolar radiofrequency in the treatment of dermatologic imperfections: clinicopathological and immunohistochemical aspects. J Drugs Dermatol. 2007 Sep;6(9):890-6. PubMed PMID: 17941360.
- 11. Elman M, Vider I, Harth Y, Gottfried V, Shemer A. Non-invasive therapy of wrinkles and lax skin using a novel multisource phase-controlled radio frequency system. J Cosmet Laser Ther. 2010 Apr;12(2):81-6. PubMed PMID: 20331345.


- 12. Sadick N, Magro C. A study evaluating the safety and efficacy of the VelaSmooth system in the treatment of cellulite. J Cosmet Laser Ther. 2007 Mar;9(1):15-20. PubMed PMID: 17506136.
- 13. Brightman L, Weiss E, Chapas AM, Karen J, Hale E, Bernstein L, Geronemus RG. Improvement in arm and post-partum abdominal and flank subcutaneous fat deposits and skin laxity using a bipolar radiofrequency, infrared, vacuum and mechanical massage device. Lasers Surg Med. 2009 Dec;41(10):791-8. PubMed PMID: 20014259.
- 14. Sadick NS, Mulholland RS. A prospective clinical study to evaluate the efficacy and safety of cellulite treatment using the combination of optical and RF energies for subcutaneous tissue heating. J Cosmet Laser Ther. 2004 Dec;6(4):187-90. PubMed PMID: 16020202
- 15. Alster TS, Lupton JR. Nonablative cutaneous remodeling using radiofrequency devices. Clin Dermatol. 2007 Sep-Oct;25(5):487-91. Review. PubMed PMID: 17870527.
- 16. Zelickson BD, Kist D, Bernstein E, Brown DB, Ksenzenko S, Burns J, Kilmer S, Mehregan D, Pope K. Histological and ultrastructural evaluation of the effects of a radiofrequency-based nonablative dermal remodeling device: a pilot study. Arch Dermatol. 2004 Feb;140(2):204-9. PubMed PMID: 14967794.
- 17. Lack EB, Rachel JD, D'Andrea L, Corres J. Relationship of energy settings and impedance in different anatomic areas using a radiofrequency device. Dermatol Surg. 2005 Dec;31(12):1668-70. PubMed PMID: 16336885.
- 18. Sadick NS. Combination radiofrequency and light energies: electro-optical synergy technology in esthetic medicine. Dermatol Surg. 2005 Sep;31(9 Pt 2):1211-7; discussion 1217. PubMed PMID: 16176773.
- 19. Clinical investigation of medical devices for human subjects Good clinical practice. ISO, 2011. 14155.


# **Appendix 1: Study Schedule**




# **Appendix 2: Pain Rating Scale**

Subjects will be instructed to rate the pain associated with RF treatment by indicating a number that best represents the overall average pain experienced using the following scale:




**Appendix 3: Fitzpatrick Skin Type Classification** 




# Appendix 4: Before and After Treatment Instructions

## **Before Treatment Instructions:**

The day before and the day of your truSculpt treatment, drink plenty of water to ensure you are well hydrated. The truSculpt treatment works best when patients have had plenty of fluids prior to treatment.

## **After Treatment Care Instructions:**

- Redness is expected and should resolve within a few hours.
- Mild swelling may occur and should go away within 72 hours.
- > Tenderness of the treatment area may persist up to 1 week.
- Avoid hot showers or baths and avoid scrubbing the treated area when bathing.
- Please call your study doctor if you experience any of the following in your treatment area:
  - Blistering
  - Bleeding
  - o Burn
  - Crusting or scabbing
  - o Pain or Tenderness, Redness or Swelling that lasts more than 72 hours
  - Nodules or lumps
- > Do not pop or un-roof blisters if they occur.
- If you need to take any over-the-counter medications for discomfort after the RF treatment, take non-aspirin pain medications, such as Tylenol or Advil.
